CLINICAL TRIAL: NCT04439539
Title: A Phase 2, Randomized, Open-label, Multicenter Study to Evaluate Efficacy, Pharmacokinetics, Safety, and Tolerability of Treatment With JNJ-73763989, Pegylated Interferon Alpha-2a, Nucleos(t)Ide Analog With or Without JNJ-56136379 in Treatment-naive Patients With HBeAg Positive Chronic Hepatitis B Virus Infection
Brief Title: A Study of JNJ-73763989, Pegylated Interferon Alpha-2a, Nucleos(t)Ide Analog (NA) With or Without JNJ-56136379 in Treatment-naive Participants With Hepatitis B e Antigen (HBeAg) Positive Chronic Hepatitis B Virus (HBV) Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108815; 73763989PAHPB2005 (Other: Janssen Research & Development, LLC); 2019-004978-26 (EudraCT Number)
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir; tenofovir alafenamide; JNJ-56136379

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Participants Enrolled Prior to Protocol Amendment 5 is in Effect (Experimental): During the Induction phase, participants will receive JNJ-73763989 subcutaneously along with JNJ-56136379 tablet orally with NA (either tenofovir disoproxil or tenofovir alafenamide tablets orally) treatment. At the start of consolidation phase, participants will be randomized to receive PegIFN-alpha-2a subcutaneously in addition to JNJ-73763989 and JNJ-56136379 with NA in arm 1 and arm 2 (without PegIFN-alpha-2a). According to predefined criteria NA treatment may be continued during the follow up (FU) phase.
  Interventions: Drug: JNJ-73763989; Drug: PegIFN-alpha-2a; Drug: Tenofovir disoproxil; Drug: Tenofovir alafenamide; Drug: JNJ-56136379
- Cohort 2: Participants Enrolled After Protocol Amendment 5 is in Effect (Experimental): Following implementation of protocol amendment- 5 and 6, all participants will receive JNJ-73763989 subcutaneously along with NA (tenofovir disoproxil tablets orally) for 36 weeks (induction phase). In the consolidation phase, participants will receive PegIFN-alpha-2a subcutaneously in addition to JNJ-73763989 and NA for 12 weeks. According to predefined criteria NA treatment may be continued during the follow up (FU) phase. JNJ-56136379 (JNJ-6379) was discontinued as per amendment 6 of the study.
  Interventions: Drug: JNJ-73763989; Drug: PegIFN-alpha-2a; Drug: Tenofovir disoproxil

INTERVENTIONS:
Drug: JNJ-73763989 — JNJ-73763989 injection will be administered subcutaneously.
  Other Names: JNJ-3989
Drug: PegIFN-alpha-2a — PegIFN-alpha-2a injection will be administered subcutaneously.
Drug: Tenofovir disoproxil — Tenofovir disoproxil film-coated tablet will be administered orally.
Drug: Tenofovir alafenamide — Tenofovir alafenamide film-coated tablet will be administered orally.
  Arms: Cohort 1: Participants Enrolled Prior to Protocol Amendment 5 is in Effect
Drug: JNJ-56136379 — JNJ-56136379 will be administered orally.
  Other Names: JNJ-6379
  Arms: Cohort 1: Participants Enrolled Prior to Protocol Amendment 5 is in Effect

SUMMARY:
The purpose of this study is to evaluate the efficacy of a treatment regimen of JNJ-73763989 + pegylated interferon alpha-2a (PegIFN-alpha-2a) + nucleos(t)ide analog (NA).

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) is a small deoxyribonucleic acid virus that specifically infects the human liver. The acute phase of infection is either followed by an immune controlled state or progresses to chronic hepatitis B. The worldwide estimated prevalence of chronic HBV infection is about 292 million people affected. Hepatitis B surface antigen (HBsAg) seroclearance is currently considered to be associated with the most thorough suppression of HBV replication (termed functional cure). With current available NA treatment strategies, rate of HBsAg seroclearance remains very low (around 3 percent [%]) even under long-term treatment. Also, with the persistently high global prevalence of HBV-associated mortality, there is a medical need for more effective finite treatment options that lead to sustained HBsAg seroclearance. JNJ-73763989 is a liver-targeted antiviral therapeutic for subcutaneous injection designed to treat chronic HBV infection via a ribonucleic acid interference (RNAi) mechanism. JNJ-56136379 is an orally administered capsid assembly modulator (CAM) that is being developed for the treatment of chronic HBV infection. The aim of the study is to evaluate the efficacy of a treatment regimen of JNJ-73763989 + PegIFN-alpha-2a + NA with or without JNJ-56136379 in participants with hepatitis B e antigen (HBeAg) positive chronic infection. The study will be conducted in 4 phases: a screening phase, an induction phase with flexible duration, a consolidation phase with or without PegIFN-α2a and a follow-up phase. Safety assessments will include Adverse Events (AEs), serious AEs of the study interventions, clinical laboratory tests, Electrocardiograms (ECGs), vital signs, and physical examinations. The study title reflects the original study design and JNJ-56136379 (JNJ-6379) was initially part of the study intervention but was discontinued as per amendment 6 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable based on physical examination, medical history, vital signs, laboratory values, and 12-lead Electrocardiogram (ECG) at screening
* Currently not treated chronic hepatitis B virus (HBV) infection with alanine transaminase (ALT) less than (<) 2* upper limit of normal (ULN) at screening and HBV deoxyribonucleic acid (DNA) greater than or equal to (>=) 20,000 international units per milliliter (IU/mL)
* Body mass index (BMI) between 18.0 and 35.0 kilogram per meter square (kg/m^2), extremes included
* Liver fibrosis stage 0-2 (Metavir) or Fibroscan less than or equal to (<=) 9 Kilopascal (kPa) at screening

Exclusion Criteria:

* Evidence of infection with hepatitis A, C, D or E virus infection or evidence of human immunodeficiency, virus type 1 (HIV-1) or HIV-2 infection at screening
* History or evidence of clinical signs or symptoms of hepatic decompensation, including but not limited to: portal hypertension, ascites, hepatic encephalopathy, esophageal varices
* Evidence of liver disease of non-HBV etiology
* Participants with a history of malignancy within 5 years before screening
* Participants who had or planned major surgery, (example, requiring general anesthesia) or who have received an organ transplant
* Contraindications to the use of PegIFN-α2a

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2024-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (47):
- United States (3):
  - Ruane Clinical Research Group Inc, Los Angeles, California
  - UPMC Center For Liver Diseases, Pittsburgh, Pennsylvania
  - Liver Institute Northwest, Seattle, Washington
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - GI Research Institute (G.I.R.I.), Vancouver, British Columbia
  - Vancouver ID Research and Care Centre Society, Vancouver, British Columbia
  - Toronto General Hospital, Toronto, Ontario
- France (7):
  - Hopital Beaujon, Clichy
  - CHU de Grenoble Hopital Albert Michallon, Grenoble
  - Hopital de La Croix Rousse, Lyon
  - CHU Nantes - Hotel Dieu, Nantes
  - CHU Hopital Saint Antoine, Paris
  - Chu Rennes Hopital Pontchaillou, Rennes
  - CHU Nancy Brabois, Vandœuvre-lès-Nancy
- Germany (4):
  - Zentrum für Infektiologie Berlin Prenzlauer Berg GmbH, Berlin
  - Universitatsklinikum Essen, Essen
  - Universitätsklinikum Johann Wolfgang Goethe- Universität Frankfurt Medizinische Klinik 1, Frankfurt
  - Medizinische Hochschule Hannover, Hanover
- Japan (5):
  - Hiroshima University Hospital, Hiroshima
  - Nara Medical University Hospital, Kashihara
  - Musashino Red Cross Hospital, Musashino
  - Nagoya City University Hospital, Nagoya
  - Yokohama City University Medical Center, Yokohama
- Russia (7):
  - Irkutsk State Medical University, Irkutsk
  - Republic Clinical Infectious Hospital n.a. AF Agafonov, Kazan'
  - St. Petersburg City Center for AIDS and Infectious Diseases Treatment and Prophylaxis, Saint Petersburg
  - Clinical Infectious Diseases Hospital n. a. S.P. Botkin, Saint Petersburg
  - Medical Company Hepatolog Ltd, Samara
  - Smolensk Regional Clinical Hospital, Smolensk
  - Stavropol State Medical University, Stavropol
- Spain (3):
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Gral. Univ. Valencia, Valencia
- Taiwan (4):
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (6):
  - Hacettepe University Hospital, Ankara
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Umraniye Training and Research Hospital, Istanbul
  - Ege University Medical of Faculty, Department of Gastroenterology, Izmir
  - Acibadem Mehmet Ali Aydinlar University, Küçükçekmece
  - Karadeniz Teknik University Medical Faculty, Trabzon
- United Kingdom (4):
  - NHS Greater Glasgow and Clyde - Gartnavel General Hospital, Glasgow
  - Glasgow Royal Infirmary, Glasgow
  - Grahame Hayton Unit, London
  - Kings College Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Kennedy PTF, Fung S, Buti M, Yilmaz G, Chuang WL, Asselah T, Kurosaki M, Jezorwski J, Klyashtornyy V, Verbinnen T, Kakuda TN, Lenz O, Guinard-Azadian C, Biermer M. Peginterferon alpha-2a add-on to siRNA JNJ-73763989 in untreated patients with HBeAg-positive chronic hepatitis B virus (HBV) infection: the phase 2 REEF-IT study. Gut. 2025 Nov 4:gutjnl-2025-336592. doi: 10.1136/gutjnl-2025-336592. Online ahead of print. PMID 41193172

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Per protocol amendment (PA) 6, all participants stopped JNJ-56136379 (JNJ-6379) treatment and switched to single-arm study design: JNJ-73763989 (JNJ-3989) plus nucleos(t)ide analog (NA; tenofovir disoproxil/tenofovir Alafenamide) plus pegylated interferon alpha-2a (PegIFN-alpha-2a). The Study had of 3 phases: induction phase (IP), consolidation phase (CP) and follow-up (FU) phase.
Pre-assignment Details: Response-guided treatment (RGT): Hepatitis B surface antigen (HBsAg) less than (<) 10 international unit per millilitre (IU/mL). Post PA 5, RGT criterion was removed. Nucleos(t)ide (NA) treatment completion criteria: HBsAg <10 IU/mL, HB envelop antigen (HBeAg)-negative, and HB virus deoxyribonucleic acid (HBV DNA) <lower limit of quantification (LLOQ) and alanine aminotransferase (ALT) <3*upper limit of normal (ULN).
Groups:
- Cohort 1: JNJ-3989 200 mg+ JNJ-6379 250 mg+ NA (245/25 mg) + PegIFN-alpha-2a 180 mcg: Prior to PA 5, participants enrolled in induction phase (IP)received JNJ-3989 200 milligrams (mg) subcutaneous (SC) injection once every 4 weeks (Q4W) + JNJ-6379 250 mg tablets orally once daily (QD) + NA (TDF 245 mg/TAF 25 mg) tablet orally QD for >=36 to <=52 weeks. Participants who met RGT criterion/reached 52 weeks were considered to complete IP and entered 12-week consolidation phase (CP) and randomized to JNJ-3989 + JNJ-6379 + NA or JNJ-3989+JNJ-6379 + NA + PegIFN-alpha-2a 180 micrograms (mcg) SC injection once weekly (QW). Post PA 5, participant who did not reach IP Week 36, started PegINF-alpha-2a at Week 36 for 12 weeks and who passed IP Week 36 and/or were randomized to CP without PegINF-alpha-2a, started pegINF-alpha-2a at their next visit. Per PA 6, JNJ-6379 treatment was stopped. Post CP Week 12, participants entered 48-week FU phase and stopped JNJ-3989+PegIFN-alpha-2a. If NA treatment completion criteria (HBsAg <10 IU/mL, HBeAg negative, and HBV DNA <LLOQ and ALT <3*ULN) was met at CP Week 12, NA was stopped at FU phase Week 2, if NA treatment completion criteria was not met, NA was continued till end of FU phase.
- Cohort 1: JNJ-3989 200 mg+ NA (245/25 mg) + PegIFNalpha-2a 180 mcg: In IP, participants (enrolled prior to PA 5) received JNJ-3989 200 mg SC injection for Q4W plus NA (tenofovir disoproxil 245 mg/tenofovir alafenamide 25 mg) tablets orally QD for >=36 to <=52 weeks. Per PA 5, the end of IP was fixed to Week 36 or to the next planned visit following implementation of PA 5. After completion of IP, all participants entered 12-week CP during which PegINF-alpha-2a 180 mcg SC injection QW was added to their treatment regimen for 12-weeks. After completion of 12-week CP, all participants entered the 48-week FU phase and stopped treatment with JNJ-3989 plus PegIFN-alpha-2a. If NA treatment completion criteria was met at CP Week 12 NA was stopped at FU Week 2, if NA treatment completion criteria was not met, NA was continued till the end of FU phase.
- Cohort 2: JNJ-3989 200 mg+ NA (245/25 mg)+ PegIFNalpha-2a 180 mcg: Participants enrolled as per PA 5 and 6 received JNJ-3989 200 mg SC injection for Q4W plus NA (tenofovir disoproxil 245 mg/tenofovir alafenamide 25 mg) tablet orally QD for 36 weeks in IP. After completion of IP, participants entered 12-week CP and received PegIFN-alpha-2a 180 mcg QW for 12-week. After completion of 12-week CP, all participants entered the 48-week FU phase and stopped treatment with JNJ-3989 plus NA plus PegIFN-alpha-2a. If NA treatment completion criteria was met at CP Week 12 NA was stopped at FU Week 2, if NA treatment completion criteria was not met NA was continued till the end of FU phase.
Period: IP:Day 1-Week 36(Post-PA5)/52(Prior-PA5)
Arm/Group | Cohort 1: JNJ-3989 200 mg+ JNJ-6379 250 mg+ NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | Cohort 1: JNJ-3989 200 mg+ NA (245/25 mg) + PegIFNalpha-2a 180 mcg | Cohort 2: JNJ-3989 200 mg+ NA (245/25 mg)+ PegIFNalpha-2a 180 mcg
Started | 27 | 8 | 19
Completed | 26 | 8 | 17
Not Completed | 1 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 2
Period: Consolidation Phase (CP):CP Week 1 to 12
Arm/Group | Cohort 1: JNJ-3989 200 mg+ JNJ-6379 250 mg+ NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | Cohort 1: JNJ-3989 200 mg+ NA (245/25 mg) + PegIFNalpha-2a 180 mcg | Cohort 2: JNJ-3989 200 mg+ NA (245/25 mg)+ PegIFNalpha-2a 180 mcg
Started | 25 (1 participant discontinued JNJ-3989 treatment due to treatment failure/relapse and moved directly to FU phase without CP.) | 7 (1 participant discontinued JNJ-3989 treatment due to treatment failure/relapse and moved directly to FU phase without CP.) | 17
Completed | 25 | 7 | 17
Not Completed | 0 | 0 | 0
Period: Follow-up (FU) Phase: FU Week 1 to 48
Arm/Group | Cohort 1: JNJ-3989 200 mg+ JNJ-6379 250 mg+ NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | Cohort 1: JNJ-3989 200 mg+ NA (245/25 mg) + PegIFNalpha-2a 180 mcg | Cohort 2: JNJ-3989 200 mg+ NA (245/25 mg)+ PegIFNalpha-2a 180 mcg
Started | 26 (1 participant moved directly to FU phase without CP.) | 8 (1 participant moved directly to FU phase without CP.) | 17
Completed | 26 | 6 | 17
Not Completed | 0 | 2 | 0
Not completed — Other | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: JNJ-3989 200 mg + JNJ-6379 250 mg+ NA (245/25 mg) + PegIFN-alpha-2a 180 mcg: Prior to PA 5, participants enrolled in induction phase (IP) received JNJ-3989 200 milligrams (mg) subcutaneous (SC) injection once every 4 weeks (Q4W) + JNJ-6379 250 mg tablets orally once daily (QD) + NA (TDF 245 mg/TAF 25 mg) tablet orally QD for >=36 to <=52 weeks. Participants who met RGT criterion/reached 52 weeks were considered to complete IP and entered 12-week consolidation phase (CP) and randomized to JNJ-3989 + JNJ-6379 + NA or JNJ-3989+JNJ-6379 + NA + PegIFN-alpha-2a 180 micrograms (mcg) SC injection once weekly (QW). Post PA 5, participant who did not reach IP Week 36, started PegINF-alpha-2a at Week 36 for 12 weeks and who passed IP Week 36 and/or were randomized to CP without PegINF-alpha-2a, started pegINF-alpha-2a at their next visit. Per PA 6, JNJ-6379 treatment was stopped. Post CP Week 12, participants entered 48-week FU phase and stopped JNJ-3989+PegIFN-alpha-2a. If NA treatment completion criteria (HBsAg <10 IU/mL, HBeAg negative, and HBV DNA <LLOQ and ALT <3*ULN). was met at CP Week 12, NA was stopped at FU phase Week 2, if NA treatment completion criteria was not met, NA was continued till end of FU phase.
- Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg: In IP, participants (enrolled prior to PA 5) received JNJ-3989 200 mg SC injection for Q4W plus NA (tenofovir disoproxil 245 mg/tenofovir alafenamide 25 mg) tablets orally QD for >=36 to <=52 weeks. Per PA 5, the end of IP was fixed to Week 36 or to the next planned visit following implementation of PA 5. After completion of IP, all participants entered 12-week CP during which PegINF-alpha-2a 180 mcg SC injection QW was added to their treatment regimen for 12-weeks. After completion of 12-week CP, all participants entered the 48-week FU phase and stopped treatment with JNJ-3989 plus PegIFN-alpha-2a. If NA treatment completion criteria was met at CP Week 12 NA was stopped at FU Week 2, if NA treatment completion criteria was not met, NA was continued till the end of FU phase.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: JNJ-3989 200 mg + JNJ-6379 250 mg+ NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | Cohort 2: JNJ-3989 200 mg+ NA (245/25 mg)+ PegIFNalpha-2a 180 mcg | Total
Number analyzed (Participants) | 27 | 8 | 19 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (9.95) | 27.3 (9.95) | 33.6 (11.15) | 33.6 (10.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 3 | 8 | 26
  Male | 12 | 5 | 11 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 26 | 8 | 18 | 52
  Unknown or Not Reported | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 13 | 3 | 14 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 4 | 7
  White | 12 | 3 | 1 | 16
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  CANADA | 3 | 0 | 4 | 7
  FRANCE | 3 | 1 | 2 | 6
  GERMANY | 1 | 0 | 1 | 2
  JAPAN | 4 | 0 | 0 | 4
  RUSSIAN FEDERATION | 7 | 2 | 1 | 10
  SPAIN | 1 | 0 | 7 | 8
  TAIWAN | 1 | 0 | 1 | 2
  TURKEY | 6 | 3 | 0 | 9
  UNITED KINGDOM | 1 | 1 | 3 | 5
  UNITED STATES | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Functional Cure: Hepatitis B Surface Antigen (HBsAg) Seroclearance at 24 Weeks After Stopping All Study Interventions at the End of Consolidation Phase (CP) and Without Restarting Nucleos(t)Ide Analog (NA) Treatment
Description: Percentage of participants with functional cure (defined as percentage of participants with HBsAg seroclearance at 24 weeks after stopping all study interventions at the end of consolidation phase and without restarting NA treatment) were reported. Seroclearance HBsAg was defined as a (quantitative) HBsAg level <lower limit of quantification (LLOQ; <0.05 international units per milliliter [IU/mL]).
Time Frame: At follow-up (FU) phase Week 24
Population: Per protocol analysis set: all randomized/enrolled participants who received at least 1 dose of CP study intervention and did not had any of the selected major protocol deviations that might affect the assessment of efficacy in terms of the primary endpoint at 24 weeks after stopping all study interventions of the CP.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: JNJ-3989 200 mg+ JNJ-6379 250 mg+ NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | Cohort 1: JNJ-3989 200 mg+ NA (245/25 mg) + PegIFNalpha-2a 180 mcg | Cohort 2: JNJ-3989 200 mg+ NA (245/25 mg)+ PegIFNalpha-2a 180 mcg
Number analyzed (Participants) | 26 | 8 | 17
percentage of participants | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Number of participants with TEAEs were reported. An adverse event (AE) was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the study intervention. Treatment-emergent AEs are all AEs with an onset on or after the first administration of study treatment or any ongoing event that worsened in severity, intensity or frequency after the first administration of study treatment.
Time Frame: IP: From Day 1 up to end of IP (up to Week 52 for Cohort 1; up to Week 36 for Cohort 2); CP: CP Week 1 up to CP Week 12 (for Cohort 1 and 2); FU phase: FU Week 1 up to FU Week 48 (up to Week 112 [Cohort 1]; up to Week 96 [Cohort 2])
Population: Safety analysis set included all participants who received at least one dose of study intervention. Participants were analyzed according to the study intervention they actually received.
Measure: Count of Participants; unit: Participants
Groups:
- IP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+ PegIFN-alpha-2a 180 mcg: Prior to PA 5, participants received JNJ-3989 200 mg SC injection for Q4W + JNJ-6379 250 mg tablets orally QD plus NA (TAD 245 mg/TAF 25 mg) tablet orally QD in IP for a RGT duration for >=36-weeks to <=52-weeks.
- IP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg: In IP, participants (enrolled prior to PA 5) received JNJ-3989 200 mg SC injection for Q4W plus NA (TAD 245 mg/TAF 25 mg) tablets orally QD in IP for >=36-weeks to <=52-weeks. Per PA 5, the end of IP was fixed to Week 36 or to the next planned visit following implementation of PA 5.
- IP: Cohort 2 : JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg: Participants enrolled as per PA 5 and 6, received JNJ-3989 200 mg SC for Q4W plus NA (TAD 250 mg/TAF 25 mg) tablet orally QD in IP for 36 weeks.
- CP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg: After completion of IP, participants entered in 12 week CP and received JNJ-3989 200 mg SC Q4W plus JNJ-6379 250 tablets QD plus NA (either TAD 250 mg or TAF 25 mg) tablet orally QD from CP Week 1 to 12 and PegIFN-alpha-2a 180 mcg SC injection was added to their treatment regimen for 12 weeks.
- CP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg; CP: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg: After completion of IP, participants entered in 12-week CP and received JNJ-3989 200 mg SC injection Q4W + NA (TDF 245 mg/TAF 25 mg) tablets orally QD from CP Week 1 to 12 and PegIFN-alpha2a 180 mcg SC QW was added to their treatment regimen for 12 weeks.
- FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg; FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg: After completion of CP, all participants entered 48-Week FU phase and stopped treatment with JNJ-3989 plus JNJ-6379 plus NA (TAD 245 mg/TAF 25 mg) plus PegIFN-alpha2a. If NA treatment completion criteria was met at CP Week 12 NA was stopped at FU Week 2, if NA treatment completion criteria was not met, NA (TAD 245 mg/TAF 25 mg) was continued till the end of FU phase.
- FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg: After completion of CP, all participants entered 48-Week FU phase and stopped treatment with JNJ-3989 plus NA (TAD 245 mg/TAF 25 mg) plus PegIFN-alpha2a. If NA treatment completion criteria was met at CP Week 12, NA treatment was stopped at FU Week 2, if NA treatment completion criteria was not met, NA (TAD 245 mg/TAF 25 mg) was continued till the end of FU phase.
Arm/Group | IP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+ PegIFN-alpha-2a 180 mcg | IP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | IP: Cohort 2 : JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 27 | 8 | 19 | 25 | 7 | 17 | 26 | 8 | 17
Participants | 22 | 8 | 15 | 22 | 7 | 13 | 17 | 5 | 11

3. Secondary Outcome: Number of Participants With Treatment Emergent Serious Adverse Events (TESAEs)
Description: Number of participants with TESAEs were reported. was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the study intervention. Treatment-emergent AEs are all AEs with an onset on or after the first administration of study treatment or any ongoing event that worsened in severity, intensity or frequency after the first administration of study treatment. A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | IP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+ PegIFN-alpha-2a 180 mcg | IP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | IP: Cohort 2 : JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 27 | 8 | 19 | 25 | 7 | 17 | 26 | 8 | 17
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

4. Secondary Outcome: Number of Participants With Worst (Grade 3 or 4) Treatment-emergent DAIDS Toxicity Grade in Clinical Laboratory Tests
Description: Clinical laboratory test parameters were Hematology: absolute lymphocyte count, absolute neutrophil count (ANC), hemoglobin, Neutrophils Band Form, Neutrophils segmented, white blood cells (WBC) decreased, ; Chemistry: alanine aminotransferase (ALT) & serum glutamic pyruvic transaminase (SGPT), aspartate aminotransferase(AST)/serum glutamic oxaloacetic transaminase (SGOT), cholesterol (fasting), creatinine Kinase, creatinine, GFR from Creatinine Adjusted for BSA, GFR from Cystatin C Adjusted for BSA, low-density lipoprotein (LDL), triglycerides (fasting); Urinalysis: glycosuria. DAIDS toxicity grades: Grade 1 (Mild), Grade 2 (Moderate), Grade 3 (Severe), Grade 4 (Potentially Life-Threatening). Number of participants with treatment-emergent DAIDS toxicity Grade 3 or 4 were reported in this outcome measure.
Time Frame: as for outcome 2
Population: Safety analysis set included all participants who received at least one dose of study intervention. Participants were analyzed according to the study intervention they actually received. Here, "n"(number analyzed) signifies number of participants analyzed at specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | IP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+ PegIFN-alpha-2a 180 mcg | IP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | IP: Cohort 2 : JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 27 | 8 | 19 | 25 | 7 | 17 | 26 | 8 | 17
Participants
  Hematology: Absolute Lymphocyte Count: Low: Grade 3: number analyzed (Participants) | 26 | 8 | 19 | 25 | 7 | 17 | 26 | 8 | 17
  Hematology: Absolute Lymphocyte Count: Low: Grade 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Hematology: Absolute Neutrophil Count: Grade 3: number analyzed (Participants) | 26 | 8 | 19 | 25 | 7 | 17 | 26 | 8 | 17
  Hematology: Absolute Neutrophil Count: Grade 3 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Hematology: Hemoglobin: Low: Grade 3: number analyzed (Participants) | 26 | 8 | 19 | 25 | 7 | 17 | 26 | 8 | 17
  Hematology: Hemoglobin: Low: Grade 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Hematology: Neutrophils Band Form: Low: Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 1
  Hematology: Neutrophils Band Form: Low: Grade 4 |  |  |  | 3 |  |  | 1 |  | 1
  Hematology: Neutrophils Segmented: Low: Grade 3: number analyzed (Participants) | 26 | 8 | 19 | 25 | 7 | 17 | 26 | 8 | 17
  Hematology: Neutrophils Segmented: Low: Grade 3 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Hematology: WBC Decreased: Low: Grade 3: number analyzed (Participants) | 26 | 8 | 19 | 25 | 7 | 17 | 26 | 8 | 17
  Hematology: WBC Decreased: Low: Grade 3 | 0 | 0 | 0 | 3 | 0 | 1 | 1 | 0 | 0
  Chemistry: ALT or SGPT: High: Grade 3: number analyzed (Participants) | 26 | 8 | 19 | 25 | 7 | 17 | 26 | 8 | 17
  Chemistry: ALT or SGPT: High: Grade 3 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
  Chemistry: AST or SGOT: High: Grade 3: number analyzed (Participants) | 26 | 8 | 19 | 25 | 7 | 17 | 26 | 8 | 17
  Chemistry: AST or SGOT: High: Grade 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Chemistry: Cholesterol (Fasting): High: Grade 3: number analyzed (Participants) | 26 | 8 | 19 | 25 | 7 | 17 | 26 | 8 | 17
  Chemistry: Cholesterol (Fasting): High: Grade 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Chemistry: Creatinine Kinase : High: Grade 3: number analyzed (Participants) | 26 | 8 | 19 | 25 | 7 | 17 | 26 | 8 | 17
  Chemistry: Creatinine Kinase : High: Grade 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Chemistry: Creatinine Kinase : High: Grade 4: number analyzed (Participants) | 26 | 8 | 19 | 25 | 7 | 17 | 26 | 8 | 17
  Chemistry: Creatinine Kinase : High: Grade 4 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Chemistry: GFR from Cr Adjusted for BSA, Low: Grade 3: number analyzed (Participants) | 26 | 8 | 19 | 25 | 7 | 17 | 26 | 8 | 17
  Chemistry: GFR from Cr Adjusted for BSA, Low: Grade 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chemistry: GFR from Cy C Adjusted for BSA, Low: Grade 3: number analyzed (Participants) | 26 | 8 | 19 | 25 | 7 | 17 | 26 | 8 | 17
  Chemistry: GFR from Cy C Adjusted for BSA, Low: Grade 3 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
  Chemistry: GFR from Cy C Adjusted for BSA, Low: Grade 4: number analyzed (Participants) | 26 | 8 | 19 | 25 | 7 | 17 | 26 | 8 | 17
  Chemistry: GFR from Cy C Adjusted for BSA, Low: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Chemistry: LDL (Fasting): High: Grade 3: number analyzed (Participants) | 26 | 8 | 19 | 25 | 7 | 17 | 26 | 8 | 17
  Chemistry: LDL (Fasting): High: Grade 3 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Chemistry: Triglycerides (Fasting): High: Grade 3: number analyzed (Participants) | 26 | 8 | 19 | 25 | 7 | 17 | 26 | 8 | 17
  Chemistry: Triglycerides (Fasting): High: Grade 3 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
  Urinalysis: Glycosuria: Grade 3: number analyzed (Participants) | 17 | 7 | 7 | 13 | 6 | 6 | 12 | 8 | 5
  Urinalysis: Glycosuria: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

5. Secondary Outcome: Number of Participants With Worst Treatment-emergent Abnormality in Electrocardiogram (ECGs)
Description: Number of participants with worst treatment-emergent abnormality in ECG were reported. Treatment-emergent abnormality was defined as the abnormalities that were worsened as compared to the abnormality at baseline; which also included the shift from abnormally high to abnormally low and vice-versa. ECG parameters included heart rate (HR; abnormally low, HR <45 beats per minute (bpm) and (abnormally high HR>=120 bpm; PR interval abnormally high >220 milliseconds (ms): QRS interval abnormally high >=120 ms; QT corrected (Fridericia QTcF) categories; borderline prolonged QTc interval <450 to <=480 ms), prolonged QTc interval <480 to <=500 ms) and pathologically prolonged QTc interval >500 ms).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | IP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+ PegIFN-alpha-2a 180 mcg | IP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | IP: Cohort 2 : JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 27 | 8 | 19 | 25 | 7 | 17 | 26 | 8 | 17
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Worst Treatment-emergent Abnormalities in Vital Signs
Description: Number of participants with worst treatment-emergent abnormalities in vital signs were reported. Treatment-emergent abnormality was defined as the abnormalities that were worsened as compared to the abnormality at baseline; which also included the shift from abnormally high to abnormally low and vice-versa. Abnormalities in vital signs included abnormal pulse rate (PR); abnormally low, <=45 bpm and abnormally high >=120 bpm; diastolic blood pressure (DBP) abnormally low <=50 mmHg, systolic blood pressure (SBP) abnormally low <=90 mmHg. Additionally, abnormal low SBP and DBP were <=50 mmHg and <+90 mmHg. Only those categories in which at least one participant had data were reported.
Time Frame: as for outcome 2
Population: Safety analysis was based on safety analysis set which included all participants who received at least one dose of study intervention and were analyzed according to the study intervention they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | IP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+ PegIFN-alpha-2a 180 mcg | IP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | IP: Cohort 2 : JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 26 | 8 | 19 | 25 | 7 | 17 | 26 | 8 | 17
Participants
  DBP: High: | 3 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 0
  SBP: Low | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0
  SBP: High | 2 | 1 | 3 | 1 | 0 | 0 | 2 | 1 | 1
  Pulse rate: High | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Clinically Important Abnormalities in Physical Examination
Description: Number of participants with clinically important treatment-emergent abnormalities in physical examination were reported.
Time Frame: as for outcome 2
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | IP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+ PegIFN-alpha-2a 180 mcg | IP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | IP: Cohort 2 : JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 27 | 8 | 19 | 25 | 7 | 17 | 26 | 8 | 17
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Percentage of Participants Who Reached HBsAg Less Than (<) 10 (International Units Per Milliliter [IU/mL]) at the End of the Induction Phase (EOI)
Description: Percentage of participants who reached HBsAg <10 IU/mL at the end induction phase were reported.
Time Frame: At IP Week 36 and EOI; anytime up to IP Week 52 for Cohort 1; up to IP Week 36 for Cohort 2
Population: Treated analysis set included all participants who received at least 1 dose of study treatment within this ISA. Here, "n"(number analyzed) signifies participants who were evaluable at specified timepoints. Data for this outcome measure were planned to be collected and analyzed for IP only.
Measure: Number; unit: percentage of participants
Groups:
- IP: Cohort 1: JNJ-3989 + NA + PegIFN-alpha-2a: In IP, participants (enrolled prior to PA5) received JNJ-3989 200 mg SC injection for Q4W plus NA (TAD 245 mg/TAF 25 mg) tablets orally QD in IP for >=36-weeks to <=52-weeks. Per PA 5 the end of IP was fixed to Week 36 or to the next planned visit following implementation of PA5.
Arm/Group | IP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+ PegIFN-alpha-2a 180 mcg | IP: Cohort 1: JNJ-3989 + NA + PegIFN-alpha-2a | IP: Cohort 2 : JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 26 | 7 | 19
percentage of participants
  IP Week 36: number analyzed (Participants) | 13 | 0 | 1
  IP Week 36 | 0 [0 to 0] |  | 10 [1 to 11]
  End of Induction phase | 15.4 [2 to 16] | 37.5 | 10.5 [1 to 11]

9. Secondary Outcome: Time to Achieve First Occurrence of HBsAg <10 IU/mL
Description: Time to achieve first occurrence of HBsAg <10 IU/mL were reported. Time to HBsAg <10 IU/mL was defined as the number of days between the date of first study treatment intake and the date of the first occurrence of HBsAg <10 IU/mL. Kaplan-Meier method was used for the estimation.
Time Frame: From Baseline (Day 1 of IP) up to Follow-up phase Week 48 (up to Week 112 [Cohort 1]; up to Week 96 [Cohort 2])
Population: Treated analysis set included all participants who received at least 1 dose of study treatment within this ISA.
Measure: Median (90% Confidence Interval); unit: weeks
Arm/Group | Cohort 1: JNJ-3989 200 mg+ JNJ-6379 250 mg+ NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | Cohort 1: JNJ-3989 200 mg+ NA (245/25 mg) + PegIFNalpha-2a 180 mcg | Cohort 2: JNJ-3989 200 mg+ NA (245/25 mg)+ PegIFNalpha-2a 180 mcg
Number analyzed (Participants) | 27 | 8 | 19
weeks | 48.1 [NA to NA] — NA indicates that upper limit and lower limit of CI was not estimable due to insufficient number of participants with events. | 84.3 [2.1 to NA] — NA indicates that upper limit of 90% CI was not estimable due to insufficient number of participants with events. | 48.3 [36.1 to NA] — NA indicates that upper limit of 90% CI was not estimable due to insufficient number of participants with events.

10. Secondary Outcome: Percentage of Participants Who Met Nucleos(t)Ide Analog (NA) Treatment Completion Criteria at the End of Consolidation Phase
Description: Percentage of participants meeting the protocol-defined NA treatment completion criteria at end of consolidation were reported. NA treatment completion criteria at CP Week 12 was defined as HBsAg <10 IU/mL; HBeAg-negative; HBV DNA <20 IU/mL, (that is, LLOQ); alanine aminotransferase(ALT) <3*ULN.
Time Frame: At CP Week 12 (for Cohort 1 and 2)
Population: Treated analysis set included all participants who received at least 1 dose of study treatment within this ISA. Here "N" (Number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | CP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 25 | 7 | 17
percentage of participants | 0 [0 to 0] | 0 [0 to 0] | 5.9 [0 to 0]

11. Secondary Outcome: FU Phase: Percentage of Participants With HBsAg Seroclearance 48 Weeks After Stopping All Study Interventions of the Consolidation Phase and Without Restarting NA Treatment During Follow up Phase
Description: Percentage of participants with HBsAg seroclearance 48 weeks after stopping all study interventions at the consolidation phase and without restarting NA treatment during follow up phase were reported. HBsAg seroclearance was defined as (quantitative) HBsAg < LLOQ (HBsAg 0.05 IU/mL).
Time Frame: FU Week 48 (up to Week 112 [Cohort 1]; up to Week 96 [Cohort 2])
Population: Treated analysis set included all participants who received at least 1 dose of study treatment within this ISA. Here "N" (Number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 26 | 6 | 17
percentage of participants | 11.5 [1 to 12] | 16.7 [1 to 17] | 11.8 [1 to 12]

12. Secondary Outcome: FU Phase: Percentage of Participants With Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) <LLOQ 48 Weeks After Stopping All Study Interventions of the Consolidation Phase and Without Restarting NA Treatment During Follow up Phase
Description: Percentage of participants with HBV DNA <LLOQ (<20 IU/mL) 48 weeks after stopping all study interventions of the consolidation phase and without restarting NA treatment during follow up phase were reported.
Time Frame: FU phase: FU Week 1 up to FU Week 48 (up to Week 112 [Cohort 1]; up to Week 96 [Cohort 2])
Population: Treated analysis set included all participants who received at least 1 dose of study treatment within this ISA. Here "N" (Number of participants analyzed) signifies the number of participants who were evaluable for this outcome measure. Here, N=0 signifies that data were not collected and analyzed for participants who stopped NA at the end of treatment.
Measure: Number; unit: percentage of participants
Arm/Group | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 0 | 0 | 1
percentage of participants |  |  | 0 [0 to 0]

13. Secondary Outcome: FU Phase: Number of Participants With Off-treatment Virologic HBV Flares During Follow up Phase
Description: Number of participants with off-treatment virologic HBV flares were reported. Virologic flare was defined as confirmed HBV DNA >peak threshold (lowest peak to qualify as virologic flare was HBV DNA >200 IU/mL) in participants who were off-treatment and had HBV DNA <LLOQ (<20 IU/mL) at the last observed time point on all study treatments. The 3 thresholds of virologic flare was 20,000 IU/mL, 2,000 IU/mL and 200 IU/mL. Confirmed means that the criteria was fulfilled at 2 or more consecutive time points or at the last observed time point. Off-treatment was defined as the time period after stopping all study treatments (including NA).
Time Frame: FU phase: FU Week 1 up to FU Week 48 (up to Week 112 [Cohort 1]; up to Week 96 [Cohort 2])
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 0 | 0 | 1
Participants |  |  | 0

14. Secondary Outcome: FU Phase: Number of Participants With Off-treatment Biochemical HBV Flares During Follow-up Phase
Description: Number of participants with off-treatment biochemical HBV flares were reported. Biochemical flare was defined as first date of 2 consecutive visits with confirmed ALT and/or AST >=3*ULN and >=3*nadir (lowest value observed up to start of flare). Confirmed means that the criteria was fulfilled at 2 or more consecutive time points or at the last observed time point. Off-treatment was defined as the time period after stopping all study treatments (including NA).
Time Frame: FU phase: FU Week 1 up to FU Week 48 (up to Week 112 [Cohort 1]; up to Week 96 [Cohort 2])
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 0 | 0 | 1
Participants |  |  | 0

15. Secondary Outcome: FU Phase: Number of Participants With On-treatment Biochemical Flares During Follow-up Phase
Description: Number of participants with on-treatment biochemical HBV flares were reported. Biochemical flare was defined as first date of 2 consecutive visits with confirmed ALT and/or AST >=3*ULN and >=3*nadir (lowest value observed up to start of flare). Confirmed means that the criteria was fulfilled at 2 or more consecutive time points or at the last observed time point. On-treatment was defined as the time period during which the participant received any of the study drugs.
Time Frame: FU phase: FU Week 1 up to FU Week 48 (up to Week 112 [Cohort 1]; up to Week 96 [Cohort 2])
Population: Treated analysis set included all participants who received at least 1 dose of study treatment within this ISA.
Measure: Count of Participants; unit: Participants
Arm/Group | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 26 | 8 | 17
Participants | 2 | 0 | 2

16. Secondary Outcome: FU Phase: Number of Participants With Off-treatment Clinical Flares During Follow-up Phase
Description: Clinical flares occurred either when a virologic flare (confirmed HBV DNA >peak threshold) & biochemical flare (ALT and/or AST >=3*ULN & >=3*nadir [lowest value observed during off-treatment period up to time point of meeting the flare criteria]) overlapped in time or when a biochemical flare started within 4 weeks following the end of a virologic flare. The HBV DNA thresholds were: 20,000 IU/mL, 2,000 IU/mL and 200 IU/mL. Confirmed means that criteria was fulfilled at 2 or more consecutive time points or at last observed time point. Off-treatment was defined as time period after stopping all study drugs (including NA). The start date of a clinical flare was minimum start date of virologic flare and biochemical flare.
Time Frame: FU phase: FU Week 1 up to FU Week 48(up to Week 112 [Cohort 1]; up to Week 96 [Cohort 2])
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 0 | 0 | 1
Participants |  |  | 0

17. Secondary Outcome: FU Phase: Percentage of Participants Who Required NA Re-treatment During Follow-Up Phase
Description: Percentage of participants who required NA re-treatment during follow-up phase were reported. A responder was defined as a participant who met the criteria for NA re-treatment at any time during follow-up, for those participants who met the NA treatment completion criteria at any time during the study and actually stopped NA treatment.
Time Frame: FU phase: FU Week 1 up to FU Week 48 (up to Week 112 [Cohort 1]; up to Week 96 [Cohort 2])
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 0 | 0 | 1
percentage of participants |  |  | 0 [0 to 0]

18. Secondary Outcome: FU Phase: Percentage of Participants Who Achieved Reduction (Sustained) in HBsAg Response (Per Definition 1) at Follow-up Week 48
Description: Percentage of participants with sustained (reduction) HBsAg response (per Definition 1) were reported. Sustained HBsAg response (definition 1) was defined as: For participants with FU Week 48 data: participants who had a >1 log10 decline from baseline in HBsAg and HBsAg <000 IU/mL at FU Week 48. For participants without FU Week 48 data: participants who had a HBsAg decline from baseline of >2 log10 at FU Week 24 or >1.5 log10 at FU Week 36 (most recent value used) and had HBsAg <1000 IU/mL at the last available timepoint.
Time Frame: At FU Week 48 (Week 112 [Cohort 1]; Week 96 [Cohort 2])
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 26 | 7 | 17
percentage of participants | 53.85 [1 to 56] | 57.1 [1 to 58] | 70.6 [1 to 80]

19. Secondary Outcome: Percentage of Participants Who Achieved Reduction (Sustained) in HBsAg Response (Per Definition 2) at Follow-up Week 48
Description: Percentage of participants with sustained (reduction) HBsAg response (per Definition 2) were reported. Sustained HBsAg response (per Definition 2) was defined as: for participants with a >1 log decline in HBsAg from baseline at last follow-up visit: Among the most recent three visits, the difference between log10 HBsAg at 2 of 3 last visit and 1 of 3 last visit was <0.2, and the difference between log10 HBsAg at 3 of 3 last visit and 1 of 3 last visit was <0.2.
Time Frame: At FU Week 48 (Week 112 [Cohort 1]; Week 96 [Cohort 2])
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 26 | 7 | 17
percentage of participants | 65.4 [1 to 67] | 42.9 [1 to 50] | 70.6 [1 to 71]

20. Secondary Outcome: Percentage of Participants Who Achieved Reduction (Sustained) in HBsAg Response (Per Definition 3) at Follow-up Week 48
Description: Percentage of participants with sustained (reduction) HBsAg response (per definition 3) were reported. Sustained HBsAg response (per Definition 3) was defined as: for participants with a >1 log decline in HBsAg from baseline at last follow-up visit: Among the most recent three visits, the difference between log10 HBsAg at 2 of 3 last visit and 1 of 3 last visit was <0.2, and the difference between log10 HBsAg at 3 of 3 last visit and 1 of 3 last visit was <0.2 and had an HBsAg <1000 IU/mL at the last available timepoint.
Time Frame: At FU Week 48 (Week 112 [Cohort 1]; Week 96 [Cohort 2])
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 26 | 7 | 17
percentage of participants | 42.3 [1 to 43] | 28.6 [1 to 30] | 52.9 [1 to 53]

21. Secondary Outcome: Percentage of Participants Who Achieved Reduction (Sustained) in HBsAg Response (Per Definition 4) at Follow-up Week 48
Description: Percentage of participants with sustained (reduction) HBsAg response per Definition 4 were reported. Sustained HBsAg response (per Definition 4) was defined as stable level, decreasing level, and increasing level. Stable level: when HBsAg change from consolidation week 12 to last available follow-up timepoint was within 0.2 log10. Decreasing level: when HBsAg change from consolidation week 12 to last available follow-up timepoint was less than -0.2 log10. Increasing level: when HBsAg change from consolidation week 12 to last available follow-up timepoint was more than 0.2 log10.
Time Frame: At FU Week 48 (Week 112 [Cohort 1]; Week 96 [Cohort 2])
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 26 | 7 | 17
percentage of participants
  Stable: within +/-0.2 log10 IU/mL | 0 [0 to 0] | 14.3 [0 to 15] | 11.8 [0 to 12]
  Decreased: <0.2 log10 IU/mL | 19.2 [0 to 20] | 14.3 [0 to 15] | 17.6 [0 to 18]
  Increased: > +0.2 log10 IU/mL | 76.9 [0 to 80] | 71.4 [0 to 72] | 70.6 [0 to 72]
  Missing | 3.9 | 0 | 0

22. Secondary Outcome: Percentage of Participants With HBsAg Seroclearance at Follow-up Week 48
Description: Percentage of Participants with HBsAg Seroclearance were reported. HBsAg seroclearance was defined as (quantitative) HBsAg level <LLOQ (<0.05 IU/mL).
Time Frame: At FU Week 48 (Week 112 [Cohort 1]; Week 96 [Cohort 2])
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 26 | 6 | 17
percentage of participants | 11.5 [1 to 12] | 16.7 [1 to 17] | 11.8 [1 to 90]

23. Secondary Outcome: Percentage of Participants With HBeAg Seroclearance at Follow-up Week 48
Description: Percentage of participants with HBeAg seroclearance were reported. HBeAg seroclearance was defined as (quantitative) HBeAg levels <LLOQ (<0.11 IU/mL).
Time Frame: At FU Week 48 (Week 112 [Cohort 1]; Week 96 [Cohort 2])
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 25 | 6 | 17
percentage of participants | 28.0 [1 to 30] | 33.3 [1 to 40] | 17.6 [1 to 18]

24. Secondary Outcome: Percentage of Participants With HBsAg Seroconversion
Description: Seroconversion of HBsAg was defined as having achieved HBsAg seroclearance (defined as quantitative HBsAg <LLOQ [<0.05 IU/mL]) and appearance of anti-HBs antibodies (defined as a baseline anti-HBs antibodies [quantitative] <LLOQ [<5 milli-international units per milliliter (mIU/mL)] and a post-baseline assessment >=LLOQ [>=5 mIU/mL]).
Time Frame: IP Week 24; CP: Week 12, FU phase: Week 48 (Week 112 [Cohort 1]; Week 96 [Cohort 2])
Population: Treated analysis set included all participants who received at least 1 dose of study treatment within this ISA. Here "N" (Number of participants analyzed) signifies participants who were evaluable for this outcome measure and "n" (number analyzed) signifies participants evaluable at specified timepoints. Also, n=0 signifies that data were not collected and analyzed as that timepoint was not applicable to the respective arm.
Measure: Number; unit: percentage of participants
Arm/Group | IP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+ PegIFN-alpha-2a 180 mcg | IP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | IP: Cohort 2 : JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 25 | 7 | 15 | 24 | 6 | 15 | 25 | 7 | 15
percentage of participants
  IP: Week 24: number analyzed (Participants) | 25 | 7 | 15 | 0 | 0 | 0 | 0 | 0 | 0
  IP: Week 24 | 0 | 0 | 0 |  |  |  |  |  |
  CP: Week 12: number analyzed (Participants) | 0 | 0 | 0 | 24 | 6 | 15 | 0 | 0 | 0
  CP: Week 12 |  |  |  | 8.3 | 33.3 | 6.7 |  |  |
  FU phase Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 25 | 0 | 15
  FU phase Week 48 |  |  |  |  |  |  | 12.0 |  | 6.7

25. Secondary Outcome: Percentage of Participants With HBeAg Seroconversion
Description: Percentage of participants with HBeAg seroconversion were reported. Seroconversion of HBeAg was defined as having achieved HBeAg seroclearance (defined as [quantitative] HBeAg <LLOQ [<0.11 IU/mL]) together with appearance of anti-HBe antibodies (defined as a baseline anti-HBe antibodies [qualitative] with a "negative" result and a post-baseline assessment with "positive" result).
Time Frame: CP: Week 12; FU phase: FU Week 48 (up to Week 112 [Cohort 1]; up to Week 96 [Cohort 2])
Population: Treated analysis set included all participants who received at least 1 dose of study treatment within this ISA. Here "N" (Number of participants analyzed) signifies participants who were evaluable for this outcome measure and "n"(number analyzed) signifies participants evaluable at specified timepoints. Data were planned to be collected and analyzed for CP and FU phase only. Here, n=0, signify that data were not collected and analyzed as that timepoint was not applicable to the respective arm.
Measure: Number; unit: percentage of participants
Arm/Group | CP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 21 | 6 | 11 | 22 | 7 | 11
percentage of participants
  CP: Week 12: number analyzed (Participants) | 21 | 6 | 11 | 0 | 0 | 0
  CP: Week 12 | 0 | 16.7 | 9.1 |  |  |
  FU phase: week 48: number analyzed (Participants) | 0 | 0 | 0 | 22 | 7 | 11
  FU phase: week 48 |  |  |  | 18.2 | 20.0 | 27.3

26. Secondary Outcome: Change From Baseline Over Time in HBsAg Levels
Description: Change from baseline over time in HBsAg levels at specified timepoints were reported
Time Frame: Baseline (Day 1 of IP), IP: Week 36; CP: Week 12; FU phase: Week 48 (Week 112 [Cohort 1]; Week 96 [Cohort 2])
Population: Treated analysis set included all participants who received at least 1 dose of study treatment within this ISA. Here "N" (Number of participants analyzed) signifies participants who were evaluable for this outcome measure and "n"(number analysed) signifies participants evaluable at specified timepoints. Here, n=0, signify that data were not collected and analyzed as that timepoint was not applicable to the respective arm.
Measure: Mean (Standard Error); unit: log10 IU/mL
Arm/Group | IP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+ PegIFN-alpha-2a 180 mcg | IP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | IP: Cohort 2 : JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 25 | 7 | 15 | 25 | 7 | 17 | 26 | 6 | 17
log10 IU/mL
  IP: Week 36: number analyzed (Participants) | 25 | 7 | 15 | 0 | 0 | 0 | 0 | 0 | 0
  IP: Week 36 | -2.78 (0.198) | -3.35 (0.417) | -2.73 (0.150) |  |  |  |  |  |
  CP: Week 12: number analyzed (Participants) | 0 | 0 | 0 | 25 | 7 | 17 | 0 | 0 | 0
  CP: Week 12 |  |  |  | -3.51 (0.275) | -4.17 (0.444) | -3.53 (0.285) |  |  |
  FU phase: Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 6 | 17
  FU phase: Week 48 |  |  |  |  |  |  | -2.41 (0.364) | -3.14 (0.747) | -2.82 (0.425)

27. Secondary Outcome: Change From Baseline Over Time in HBeAg Levels
Description: Change from baseline over time in HBsAg levels at specified timepoints were reported.
Time Frame: Baseline (Day 1 of IP), IP: Week 36; CP: Week 12; FU phase: Week 48 (Week 112 [Cohort 1]; Week 96 [Cohort 2])
Population: as for outcome 26
Measure: Mean (Standard Error); unit: log10 IU/mL
Arm/Group | IP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+ PegIFN-alpha-2a 180 mcg | IP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | IP: Cohort 2 : JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 24 | 7 | 15 | 24 | 7 | 17 | 25 | 6 | 17
log10 IU/mL
  IP: Week 36: number analyzed (Participants) | 24 | 7 | 15 | 0 | 0 | 0 | 0 | 0 | 0
  IP: Week 36 | -1.78 (0.103) | -1.77 (0.151) | -1.49 (0.141) |  |  |  |  |  |
  CP: Week 12: number analyzed (Participants) | 0 | 0 | 0 | 24 | 7 | 17 | 0 | 0 | 0
  CP: Week 12 |  |  |  | -2.14 (0.146) | -2.39 (0.162) | -2.22 (0.234) |  |  |
  FU phase: Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 25 | 6 | 17
  FU phase: Week 48 |  |  |  |  |  |  | -2.45 (0.243) | -2.59 (0.508) | -2.47 (0.278)

28. Secondary Outcome: Change From Baseline Over Time in HBV DNA Levels
Description: Change from baseline over time in HBV DNA Levels at Specified Timepoints were reported.
Time Frame: Baseline (Day 1 of IP), IP: Week 36; CP: Week 12; FU phase: Week 48 (Week 112 [Cohort 1]; Week 96 [Cohort 2])
Population: as for outcome 26
Measure: Mean (Standard Error); unit: log10 IU/mL
Arm/Group | IP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+ PegIFN-alpha-2a 180 mcg | IP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | IP: Cohort 2 : JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 25 | 7 | 15 | 25 | 6 | 17 | 26 | 6 | 17
log10 IU/mL
  IP: Week 36: number analyzed (Participants) | 25 | 7 | 15 | 0 | 0 | 0 | 0 | 0 | 0
  IP: Week 36 | -6.36 (0.218) | -6.08 (0.202) | -6.26 (0.231) |  |  |  |  |  |
  CP: Week 12: number analyzed (Participants) | 0 | 0 | 0 | 25 | 6 | 17 | 0 | 0 | 0
  CP: Week 12 |  |  |  | -6.29 (0.205) | -6.30 (0.350) | -6.07 (0.269) |  |  |
  FU phase: Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 6 | 17
  FU phase: Week 48 |  |  |  |  |  |  | -6.79 (0.203) | -5.95 (0.563) | -6.70 (0.257)

29. Secondary Outcome: Time to Achieve First HBsAg Seroclearance
Description: Time to achieve first HBsAg seroclearance (defined as quantitative HBsAg <LLOQ; HBsAg <0.05 IU/mL) were reported. Time to HBsAg seroclearance was defined as the number of days between the date of first study intervention intake and the date of the first occurrence of HBsAg seroclearance. Kaplan-Meier method was used for the estimation.
Time Frame: From Baseline (Day 1 of IP) to Follow-up Week 48 (up to Week 112 [Cohort 1]; up to Week 96 [Cohort 2])
Population: Treated analysis set included all participants who received at least 1 dose of study treatment within this ISA. Here "N" (Number of participants analyzed) signifies participants who were evaluable for this endpoint. Per planned analysis, data for this outcome measure was analyzed per pooled cohorts only.
Measure: Median (90% Confidence Interval); unit: weeks
Arm/Group | Cohort 1: JNJ-3989 200 mg+ JNJ-6379 250 mg+ NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | Cohort 1: JNJ-3989 200 mg+ NA (245/25 mg) + PegIFNalpha-2a 180 mcg | Cohort 2: JNJ-3989 200 mg+ NA (245/25 mg)+ PegIFNalpha-2a 180 mcg
Number analyzed (Participants) | 27 | 8 | 19
weeks | NA [NA to NA] — NA indicates that median [90% CI] data were not estimable due to insufficient number of participants with events. | NA [6.1 to NA] — NA indicates that median [90% CI] data were not estimable due to insufficient number of participants with events. | NA [NA to NA] — NA indicates that median [90% CI] data were not estimable due to insufficient number of participants with events.

30. Secondary Outcome: Time to Achieve First HBeAg Seroclearance
Description: Time to achieve first occurrence of HBeAg seroclearance (HBeAg <LLOQ [<0.11 IU/mL]) were reported. Time to first occurrence of the HBeAg seroclearance was defined as the number of days between the date of first study intervention intake and the date of the first occurrence of the HBeAg seroclearance.
Time Frame: From Baseline (Day 1 of IP) to Follow-up Week 48 (up to Week 112 [Cohort 1]; up to Week 96 [Cohort 2])
Population: Treated analysis set included all participants who received at least 1 dose of study treatment within this ISA. Here "N" (Number of participants analyzed) signifies participants who were evaluable for this outcome measure. Per planned analysis, data for this outcome measure was analyzed per pooled cohorts only.
Measure: Median (90% Confidence Interval); unit: weeks
Arm/Group | Cohort 1: JNJ-3989 200 mg+ JNJ-6379 250 mg+ NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | Cohort 1: JNJ-3989 200 mg+ NA (245/25 mg) + PegIFNalpha-2a 180 mcg | Cohort 2: JNJ-3989 200 mg+ NA (245/25 mg)+ PegIFNalpha-2a 180 mcg
Number analyzed (Participants) | 27 | 8 | 19
weeks | 112 [96.1 to NA] — NA indicates that upper interval of CI data were not estimable due to insufficient number of participants with events. | 100.3 [48.0 to NA] — NA indicates that upper interval of CI data were not estimable due to insufficient number of participants with events. | NA [59.1 to NA] — NA indicates that Median and upper interval of CI data were not estimable due to insufficient number of participants with events.

31. Secondary Outcome: Time to Achieve First HBV DNA <LLOQ
Description: Time to achieve first occurrence of HBV DNA < LLOQ (<20 IU/mL) were reported. Time to first occurrence of the HBV DNA < LLOQ was defined as the number of days between the date of first study intervention intake and the date of the first occurrence of the HBV DNA < LLOQ.
Time Frame: From Baseline (Day 1 of IP) to Follow-up Week 48 (up to Week 112 [Cohort 1]; up to Week 96 [Cohort 2])
Population: as for outcome 30
Measure: Median (90% Confidence Interval); unit: weeks
Arm/Group | Cohort 1: JNJ-3989 200 mg+ JNJ-6379 250 mg+ NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | Cohort 1: JNJ-3989 200 mg+ NA (245/25 mg) + PegIFNalpha-2a 180 mcg | Cohort 2: JNJ-3989 200 mg+ NA (245/25 mg)+ PegIFNalpha-2a 180 mcg
Number analyzed (Participants) | 27 | 8 | 19
weeks | 35.9 [28.1 to 52.1] | 53.3 [12.1 to NA] — NA indicates that lower interval of CI data were not estimable due to insufficient number of participants with events. | 38.1 [24.1 to 50.1]

32. Secondary Outcome: Percentage of Participants With HBeAg Levels Below Different Cut-offs
Description: Percentage of participants with HBeAg levels below different cut-offs were reported. The cut-offs for HBeAg levels were : <LLOQ (<0.11 IU/mL), < 1 IU/mL, < 10 IU/mL, <100 IU/mL
Time Frame: IP: Week 36, CP: Week 12; FU phase: Week 48 (Week 112 [Cohort 1]; Week 96 [Cohort 2])
Population: Treated analysis set included all participants who received at least 1 dose of study treatment within this ISA.Here "N" (Number of participants analyzed) signifies participants who were evaluable for this outcome measure and "n"(number analysed) signifies participants evaluable at specified timepoints. Here, n=0, signify that data were not collected and analyzed as that timepoint was not applicable to the respective arm.
Measure: Number; unit: percentage of participants
Arm/Group | IP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+ PegIFN-alpha-2a 180 mcg | IP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | IP: Cohort 2 : JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 24 | 7 | 15 | 24 | 7 | 17 | 25 | 6 | 17
percentage of participants
  IP Week 36: <0.11 IU/mL: number analyzed (Participants) | 24 | 7 | 15 | 0 | 0 | 0 | 0 | 0 | 0
  IP Week 36: <0.11 IU/mL | 12.5 | 0 | 0 |  |  |  |  |  |
  IP Week 36: <1 IU/mL: number analyzed (Participants) | 24 | 7 | 15 | 0 | 0 | 0 | 0 | 0 | 0
  IP Week 36: <1 IU/mL | 20.8 | 14.3 | 20.0 |  |  |  |  |  |
  IP Week 36: <10 IU/mL: number analyzed (Participants) | 24 | 7 | 15 | 0 | 0 | 0 | 0 | 0 | 0
  IP Week 36: <10 IU/mL | 54.2 | 71.4 | 46.7 |  |  |  |  |  |
  IP Week 36: <100 IU/mL: number analyzed (Participants) | 24 | 7 | 15 | 0 | 0 | 0 | 0 | 0 | 0
  IP Week 36: <100 IU/mL | 91.7 | 100.0 | 86.7 |  |  |  |  |  |
  CP Week 12: <0.11 IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 24 | 7 | 17 | 0 | 0 | 0
  CP Week 12: <0.11 IU/mL |  |  |  | 12.5 | 14.3 | 17.6 |  |  |
  CP Week 12: <1 IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 24 | 7 | 17 | 0 | 0 | 0
  CP Week 12: <1 IU/mL |  |  |  | 37.5 | 14.3 | 47.1 |  |  |
  CP Week 12: <10 IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 24 | 7 | 17 | 0 | 0 | 0
  CP Week 12: <10 IU/mL |  |  |  | 75.0 | 100.0 | 76.5 |  |  |
  CP Week 12: <100 IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 23 | 7 | 17 | 0 | 0 | 0
  CP Week 12: <100 IU/mL |  |  |  | 95.8 | 100.0 | 94.1 |  |  |
  FU Week 48: <0.11 IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 25 | 6 | 17
  FU Week 48: <0.11 IU/mL |  |  |  |  |  |  | 28.0 | 33.3 | 17.6
  FU Week 48: <1 IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 25 | 6 | 17
  FU Week 48: <1 IU/mL |  |  |  |  |  |  | 44.0 | 50.0 | 52.9
  FU Week 48: <10 IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 25 | 6 | 17
  FU Week 48: <10 IU/mL |  |  |  |  |  |  | 80.0 | 83.3 | 76.5
  FU Week 48: <100IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 25 | 6 | 17
  FU Week 48: <100IU/mL |  |  |  |  |  |  | 96.0 | 100 | 100

33. Secondary Outcome: Percentage of Participants With HBsAg Levels Below Different Cut-offs
Description: Percentage of participants with HBsAg levels below different cut-offs were reported. The cut-offs for HBsAg level were: <LLOQ (<0.05 IU/mL), <1 IU/mL, <10 IU/mL, <100 IU/mL, <1000 IU/mL.
Time Frame: IP: Week 36, CP: Week 12; FU phase: Week 48 (Week 112 [Cohort 1]; Week 96 [Cohort 2])
Population: as for outcome 32
Measure: Number; unit: percentage of participants
Arm/Group | IP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+ PegIFN-alpha-2a 180 mcg | IP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | IP: Cohort 2 : JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 25 | 7 | 15 | 25 | 7 | 17 | 26 | 6 | 17
percentage of participants
  IP Week 36: <0.05 IU/mL: number analyzed (Participants) | 25 | 7 | 15 | 0 | 0 | 0 | 0 | 0 | 0
  IP Week 36: <0.05 IU/mL | 0 | 14.3 | 0 |  |  |  |  |  |
  IP Week 36: <1 IU/mL: number analyzed (Participants) | 25 | 7 | 15 | 0 | 0 | 0 | 0 | 0 | 0
  IP Week 36: <1 IU/mL | 4.0 | 28.6 | 0 |  |  |  |  |  |
  IP Week 36: <10 IU/mL: number analyzed (Participants) | 25 | 7 | 15 | 0 | 0 | 0 | 0 | 0 | 0
  IP Week 36: <10 IU/mL | 24.0 | 42.9 | 13.3 |  |  |  |  |  |
  IP Week 36: <100 IU/mL: number analyzed (Participants) | 25 | 7 | 15 | 0 | 0 | 0 | 0 | 0 | 0
  IP Week 36: <100 IU/mL | 40.0 | 42.9 | 66.7 |  |  |  |  |  |
  IP Week 36: <1000 IU/mL: number analyzed (Participants) | 25 | 7 | 15 | 0 | 0 | 0 | 0 | 0 | 0
  IP Week 36: <1000 IU/mL | 88.0 | 100.0 | 86.7 |  |  |  |  |  |
  CP Week 12: <0.05 IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 25 | 7 | 17 | 0 | 0 | 0
  CP Week 12: <0.05 IU/mL |  |  |  | 8.0 | 42.9 | 5.9 |  |  |
  CP Week 12: <1 IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 25 | 7 | 17 | 0 | 0 | 0
  CP Week 12: <1 IU/mL |  |  |  | 20.0 | 42.9 | 23.5 |  |  |
  CP Week 12: <10 IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 25 | 7 | 17 | 0 | 0 | 0
  CP Week 12: <10 IU/mL |  |  |  | 40.0 | 42.9 | 47.1 |  |  |
  CP Week 12: <100 IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 25 | 7 | 17 | 0 | 0 | 0
  CP Week 12: <100 IU/mL |  |  |  | 60.0 | 71.4 | 76.5 |  |  |
  CP Week 12: <1000 IU0/mL: number analyzed (Participants) | 0 | 0 | 0 | 25 | 7 | 17 | 0 | 0 | 0
  CP Week 12: <1000 IU0/mL |  |  |  | 100.0 | 100.0 | 94.1 |  |  |
  FU Week 48: <0.05 IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 6 | 17
  FU Week 48: <0.05 IU/mL |  |  |  |  |  |  | 11.5 | 16.7 | 11.8
  FU Week 48: <1 IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 6 | 17
  FU Week 48: <1 IU/mL |  |  |  |  |  |  | 11.5 | 33.3 | 17.6
  FU Week 48: <10 IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 6 | 17
  FU Week 48: <10 IU/mL |  |  |  |  |  |  | 19.2 | 50.0 | 29.4
  FU Week 48: <100 IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 6 | 17
  FU Week 48: <100 IU/mL |  |  |  |  |  |  | 26.9 | 50.0 | 47.1
  FU Week 48: <1000 IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 6 | 17
  FU Week 48: <1000 IU/mL |  |  |  |  |  |  | 57.7 | 66.7 | 76.5

34. Secondary Outcome: Percentage of Participants With HBV DNA Levels Below Different Cut-offs
Description: Percentage of participants with HBV DNA levels below cut-offs were reported. The cut-offs for HBV DNA were as follows: <LLOQ (<20 IU/mL) for target detected and not detected, < LLOQ for target not detected , and < LLOQ for target detected, <60 IU/mL, <100 IU/mL, <200 IU/mL, <1000 IU/mL, <2000 IU/mL, <20000 IU/mL.
Time Frame: IP: Week 36; CP: Week 12; FU phase: Week 48 (Week 112 [Cohort 1]; Week 96 [Cohort 2])
Population: Treated analysis set included all participants who received at least 1 dose of study treatment within this ISA. Here "N" (Number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure and "n"(number of participants analyzed) signifies participants analyzed at specified categories. Here, n=0, signify that data were not collected and analyzed as that timepoint was not applicable to the respective arm.
Measure: Number; unit: percentage of participants
Arm/Group | IP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+ PegIFN-alpha-2a 180 mcg | IP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | IP: Cohort 2 : JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 25 | 7 | 15 | 25 | 6 | 17 | 26 | 6 | 17
percentage of participants
  IP Week 36:<LLOQ target detected and not detected: number analyzed (Participants) | 25 | 7 | 15 | 0 | 0 | 0 | 0 | 0 | 0
  IP Week 36:<LLOQ target detected and not detected | 52.0 | 28.6 | 40.0 |  |  |  |  |  |
  IP Week 36:<LLOQ for target not detected: number analyzed (Participants) | 25 | 7 | 15 | 0 | 0 | 0 | 0 | 0 | 0
  IP Week 36:<LLOQ for target not detected | 8.0 | 0 | 6.7 |  |  |  |  |  |
  IP Week 36:<LLOQ for target detected: number analyzed (Participants) | 25 | 7 | 15 | 0 | 0 | 0 | 0 | 0 | 0
  IP Week 36:<LLOQ for target detected | 44.0 | 28.6 | 33.3 |  |  |  |  |  |
  IP Week 36:<60 IU/mL: number analyzed (Participants) | 25 | 7 | 15 | 0 | 0 | 0 | 0 | 0 | 0
  IP Week 36:<60 IU/mL | 72.0 | 57.1 | 73.3 |  |  |  |  |  |
  IP Week 36:<100 IU/mL: number analyzed (Participants) | 25 | 7 | 15 | 0 | 0 | 0 | 0 | 0 | 0
  IP Week 36:<100 IU/mL | 88.0 | 57.1 | 80.0 |  |  |  |  |  |
  IP Week 36:<200 IU/mL: number analyzed (Participants) | 25 | 7 | 15 | 0 | 0 | 0 | 0 | 0 | 0
  IP Week 36:<200 IU/mL | 92.0 | 71.4 | 86.7 |  |  |  |  |  |
  IP Week 36:<1000 IU/mL: number analyzed (Participants) | 25 | 7 | 15 | 0 | 0 | 0 | 0 | 0 | 0
  IP Week 36:<1000 IU/mL | 100.0 | 100.0 | 100.0 |  |  |  |  |  |
  IP Week 36:<2000 IU/mL: number analyzed (Participants) | 25 | 7 | 15 | 0 | 0 | 0 | 0 | 0 | 0
  IP Week 36:<2000 IU/mL | 100.0 | 100.0 | 100.0 |  |  |  |  |  |
  IP Week 36:<20000 IU/mL: number analyzed (Participants) | 25 | 7 | 15 | 0 | 0 | 0 | 0 | 0 | 0
  IP Week 36:<20000 IU/mL | 100.0 | 100.0 | 100.0 |  |  |  |  |  |
  CP Week 12:<LLOQ: target detected and not detected: number analyzed (Participants) | 0 | 0 | 0 | 25 | 6 | 17 | 0 | 0 | 0
  CP Week 12:<LLOQ: target detected and not detected |  |  |  | 32.0 | 33.3 | 29.4 |  |  |
  CP Week 12:<LLOQ for target not detected: number analyzed (Participants) | 0 | 0 | 0 | 25 | 6 | 17 | 0 | 0 | 0
  CP Week 12:<LLOQ for target not detected |  |  |  | 0 | 0 | 0 |  |  |
  CP Week 12:<LLOQ for target detected: number analyzed (Participants) | 0 | 0 | 0 | 25 | 6 | 17 | 0 | 0 | 0
  CP Week 12:<LLOQ for target detected |  |  |  | 32.0 | 33.3 | 29.4 |  |  |
  CP Week 12:<60 IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 25 | 6 | 17 | 0 | 0 | 0
  CP Week 12:<60 IU/mL |  |  |  | 76.0 | 50.0 | 58.8 |  |  |
  CP Week 12:<100 IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 25 | 6 | 17 | 0 | 0 | 0
  CP Week 12:<100 IU/mL |  |  |  | 92.0 | 83.3 | 64.7 |  |  |
  CP Week 12:<200 IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 25 | 6 | 17 | 0 | 0 | 0
  CP Week 12:<200 IU/mL |  |  |  | 96.0 | 83.3 | 82.4 |  |  |
  CP Week 12:<1000 IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 25 | 6 | 17 | 0 | 0 | 0
  CP Week 12:<1000 IU/mL |  |  |  | 100.0 | 100.0 | 94.1 |  |  |
  CP Week 12:<2000 IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 25 | 6 | 17 | 0 | 0 | 0
  CP Week 12:<2000 IU/mL |  |  |  | 100.0 | 100.0 | 100.0 |  |  |
  CP Week 12:<20000 IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 25 | 6 | 17 | 0 | 0 | 0
  CP Week 12:<20000 IU/mL |  |  |  | 100.0 | 100.0 | 100.0 |  |  |
  FU Week 48:<LLOQ target detected and not detected: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 6 | 17
  FU Week 48:<LLOQ target detected and not detected |  |  |  |  |  |  | 84.6 | 50.0 | 88.2
  FU Week 48: <LLOQ for target not detected: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 6 | 17
  FU Week 48: <LLOQ for target not detected |  |  |  |  |  |  | 34.6 | 16.7 | 17.6
  FU Week 48:<LLOQ for target detected: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 6 | 17
  FU Week 48:<LLOQ for target detected |  |  |  |  |  |  | 50.0 | 33.3 | 70.6
  FU Week 48:<60 IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 6 | 17
  FU Week 48:<60 IU/mL |  |  |  |  |  |  | 92.3 | 50.0 | 94.1
  FU Week 48:<100 IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 6 | 17
  FU Week 48:<100 IU/mL |  |  |  |  |  |  | 100.0 | 66.7 | 100.0
  FU Week 48:<200 IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 6 | 17
  FU Week 48:<200 IU/mL |  |  |  |  |  |  | 100.0 | 83.3 | 100.0
  FU Week 48:<1000 IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 6 | 17
  FU Week 48:<1000 IU/mL |  |  |  |  |  |  | 100.0 | 83.3 | 100.0
  FU Week 48:<2000 IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 6 | 17
  FU Week 48:<2000 IU/mL |  |  |  |  |  |  | 100.0 | 83.3 | 100.0
  FU Week 48:<20000 IU/mL: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 6 | 17
  FU Week 48:<20000 IU/mL |  |  |  |  |  |  | 100.0 | 100.0 | 100.0

35. Secondary Outcome: Percentage of Participants With Virologic Breakthrough
Description: Percentage of participants with virologic breakthrough on treatment were reported. Virological breakthrough was defined as confirmed on-treatment HBV DNA increase by >1 log10 IU/mL from nadir level (lowest level reached during treatment) in participants who did not have on-treatment HBV DNA level < LLOQ (<20 IU/mL) or confirmed on-treatment HBV DNA level >200 IU/mL in participants who had on-treatment HBV DNA level <LLOQ of the HBV DNA assay. Confirmed HBV DNA increase/level means that the criterion was fulfilled at 2 or more consecutive time points or at the last observed on-treatment time point.
Time Frame: as for outcome 2
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | IP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+ PegIFN-alpha-2a 180 mcg | IP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | IP: Cohort 2 : JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | CP: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 27 | 8 | 19 | 25 | 7 | 17 | 26 | 7 | 17
percentage of participants | 3.7 | 12.5 | 0 | 0 | 0 | 0 | 0 | 50.0 | 0

36. Secondary Outcome: Percentage of Participants Who Reached HBV DNA Undetectability After Re-start of NA Treatment During Follow-up
Description: Percentage of participants who reached HBV DNA undetectability after re-start of NA treatment during follow-up were reported. Undetectability of HBV DNA was defined as HBV DNA<LLOQ that is <20 IU/mL.
Time Frame: FU phase: FU Week 1 up to FU Week 48 (up to Week 112 [Cohort 1]; up to Week 96 [Cohort 2])
Population: Treated analysis set included all participants who received at least 1 dose of study treatment within this ISA. Here N=0 signifies that data could not be analyzed due to insufficient number of participants with events.
Measure: Number; unit: percentage of participants
Arm/Group | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFN-alpha-2a 180 mcg
Number analyzed (Participants) | 27 | 8 | 19
percentage of participants | 0 | 0 | 0

37. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of JNJ-73763989 (Molecules: JNJ-73763976 [JNJ3976], JNJ-73763924 [JNJ-3924])
Description: Cmax of JNJ-73763989 (molecules: JNJ-73763976 [JNJ3976], JNJ-73763924 [JNJ-3924]) were reported. Noncompartmental analysis were conducted to analyze Cmax JNJ-73763989 and its molecules
Time Frame: IP : Predose (0 hour), post dose on 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10 and 24 hours on IP Week 24; CP: Predose (0 hour), post dose on 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10 and 24 hours on CP Week 8
Population: Pharmacokinetics analysis set (PK): included participants who had received at least 1 dose of any of the study interventions and had at least 1 valid blood sample drawn for PK analysis. Data for this outcome measure was planned to be collected and analyzed as pooled cohort in induction phase and consolidation phase only.
Measure: Mean (Standard Deviation); unit: nanogram per milliliters (ng/mL)
Groups:
- Induction Phase: Prior PA 5, participants received JNJ-3989 200 mg SC injection for Q4W + JNJ-6379 250 mg tablets orally QD plus NA (TAD 245 mg/TAF 25 mg) tablet orally QD for >=36-weeks to <=52-weeks. Participants who met RGT criterion/reached 52 weeks were considered to complete IP and entered 12-week CP and randomized to JNJ-3989 + JNJ-6379 + NA or JNJ-3989+JNJ-6379 + NA + PegIFN-alpha-2a 180 mcg SC injection QW. In IP, participants (enrolled prior to PA 5) received JNJ-3989 200 mg SC injection for Q4W plus NA (TAD 245 mg/TAF 25 mg) tablets orally QD for >=36 to <=52 weeks. Per PA 5 the end of IP was fixed to Week 36 or to the next planned visit following implementation of PA 5. Participants enrolled as per PA 5 and 6, received JNJ-3989 200 mg SC for Q4W plus NA (either tenofovir disoproxil 250 mg or 25 mg tenofovir alafenamide) tablet orally QD for 36 weeks in IP. Post PA 5, participant not reached IP Week 36, started PegINF-alpha-2a at Week 36 for 12 weeks and who passed IP Week 36 and/or were randomized to CP without PegINF-alpha-2a, started pegINF-alpha-2a at their next visit.
- Consolidation Phase: After completion of IP, participants entered the 12 weeks CP and received JNJ-3989 200 mg SC Q4W plus JNJ-6379 250 tablets QD plus NA (either TDF 245 mg/TAF 25 mg) tablet orally QD plus PegIFN-alpha-2a 180 mcg SC QW. At the end of the CP, all participants entered the 48-weeks follow-up (FU) phase and stopped treatment with JNJ-3989 plus JNJ-6379 plus NA plus PegIFN-alpha-2a.If NA treatment completion criteria was met at CP Week 12, NA was stopped at FU phase Week 2, if not met, NA was continued till end of FU phase.If NA treatment completion criteria was met at CP Week 12, NA was stopped at FU phase Week 2, if not met, NA was continued till end of FU phase.
Arm/Group | Induction Phase | Consolidation Phase
Number analyzed (Participants) | 8 | 6
nanogram per milliliters (ng/mL)
  JNJ-73763976 | 1376 (1266) | 700 (227)
  JNJ-73763924 | 279 (308) | 135 (39.9)

38. Secondary Outcome: Time to Reach the Maximum Observed Plasma Concentration (Tmax) of JNJ-73763989 (Molecules: JNJ-73763976 [JNJ3976], JNJ-73763924 [JNJ-3924])
Description: Time to reach the maximum observed plasma concentration (tmax) of JNJ-73763989 (molecules: JNJ-73763976 [JNJ3976], JNJ-73763924 [JNJ-3924]) were reported. Non-compartmental analysis were conducted to analyze tmax of JNJ-73763989 and its molecules.
Time Frame: as for outcome 37
Population: Pharmacokinetics analysis set (PK): included participants who have received at least 1 dose of any of the study interventions and had at least 1 valid blood sample drawn for PK analysis. Data for this endpoint was planned to be collected and analyzed as pooled cohort in induction phase and consolidation phase only.
Measure: Median (Full Range); unit: hour
Arm/Group | Induction Phase | Consolidation Phase
Number analyzed (Participants) | 8 | 6
hour
  JNJ-73763976 | 5.53 [2.50 to 6.00] | 3.99 [2.98 to 6.00]
  JNJ-73763924 | 4.00 [0.50 to 5.73] | 2.99 [1.00 to 4.00]

39. Secondary Outcome: Plasma Concentration 24 Hours After Administration (C24h) of JNJ-73763989 (Molecules: JNJ-73763976 [JNJ3976], JNJ-73763924 [JNJ-3924])
Description: Plasma concentration 24 hours after administration (C24h) of JNJ-73763989 (molecules: JNJ-73763976 [JNJ3976], JNJ-73763924 [JNJ-3924]) were reported. Non-compartmental analysis were conducted to analyze C24h of JNJ-73763989 and its molecules.
Time Frame: IP: 24 hours post dose on Week 24 visit; CP: 24 hours post dose on Week 8 visit
Population: Pharmacokinetics analysis set (PK): included participants who have received at least 1 dose of any of the study interventions and had at least 1 valid blood sample drawn for PK analysis. Here "N" (Number of participants analysed) signifies the number of participants that were evaluable for this outcome measure. Data for this endpoint was planned to be collected and analyzed as pooled cohort in induction phase and consolidation phase only.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Induction Phase | Consolidation Phase
Number analyzed (Participants) | 7 | 6
ng/mL
  JNJ-73763976 | 315 (213) | 381 (155)
  JNJ-73763924 | 36.9 (27.9) | 54.7 (25.0)

40. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to 24 Hours [AUC (0- 24 Hours)] of JNJ-73763989 (Molecules: JNJ-73763976 [JNJ3976], JNJ-73763924 [JNJ-3924])
Description: Area under the plasma concentration-time curve from time zero to 24hours (AUC0 to 24h) of JNJ-73763989 (molecules:JNJ-73763976 [JNJ3976], JNJ-73763924 [JNJ-3924]) were reported. Non-compartmental analysis were conducted toanalyze AUC0 to 24h of JNJ-73763989 and its molecules.
Time Frame: IP: 24 hours post dose on Week 24 visit; CP: 24 hours post dose on Week 8 visit
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: nanograms*hour per milliliters (ng*h/mL)
Arm/Group | Induction Phase | Consolidation Phase
Number analyzed (Participants) | 7 | 6
nanograms*hour per milliliters (ng*h/mL)
  JNJ-73763976 | 19109 (12482) | 12219 (3499)
  JNJ-73763924 | 3089 (1964) | 2117 (639)

ADVERSE EVENTS:
Time Frame: IP: From Day 1 up to end of IP (up to Week 52 for Cohort 1; up to Week 36 for Cohort 2); CP: CP Week 1 up to CP Week 12 (for Cohort 1 and 2); FU phase: FU Week 1 up to FU Week 48 (up to Week 112 [Cohort 1]; up to Week 96 [Cohort 2])
Description: Safety analysis was based on safety analysis set which included all participants who received at least one dose of study intervention and were analyzed according to the study intervention they actually received.
Groups:
- IP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFNalpha- 2a 180 mcg: In IP, participants (enrolled prior to PA 5) received JNJ-3989 200 mg SC injection for Q4W plus NA (TAD 245 mg/TAF 25 mg) tablets orally QD in IP for >=36-weeks to <=52-weeks. Per PA 5 the end of IP was fixed to Week 36 or to the next planned visit following implementation of PA 5.
- IP: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFNalpha- 2a 180 mcg: Participants enrolled as per PA 5 and 6, received JNJ-3989 200 mg SC for Q4W plus NA (TAD 250 mg/TAF 25 mg) tablet orally QD in IP for 36 weeks.
- CP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFNalpha- 2a 180 mcg; CP: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFNalpha- 2a 180 mcg: After completion of IP, participants entered in 12-week CP and received JNJ-3989 200 mg SC injection Q4W + NA (TDF 245 mg/TAF 25 mg) tablets orally QD from CP Week 1 to 12 and PegIFN-alpha2a 180 mcg SC QW was added to their treatment regimen for 12 weeks.
- FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFNalpha- 2a 180 mcg: After completion of CP, all participants entered 48-Week FU phase and stopped treatment with JNJ-3989 plus JNJ-6379 plus NA (TAD 245 mg/TAF 25 mg) plus PegIFN-alpha2a. If NA treatment completion criteria was met at CP Week 12 NA was stopped at FU W2, if NA treatment completion criteria was not met, NA (TAD 245 mg/TAF 25 mg) was continued till the end of FU phase.
- FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFNalpha- 2a 180 mcg: After completion of CP, all participants entered 48-Week FU phase and stopped treatment with JNJ-3989 plus NA (TAD 245 mg/TAF 25 mg) plus PegIFN-alpha2a. If NA treatment completion criteria was met at CP Week 12, NA treatment was stopped at FU Week 2, if NA treatment completion criteria was not met, NA (TAD 245 mg/TAF 25 mg) was continued till the end of FU phase.
Arm/Group | IP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+ PegIFN-alpha-2a 180 mcg | IP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFNalpha- 2a 180 mcg | IP: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFNalpha- 2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | CP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFNalpha- 2a 180 mcg | CP: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFNalpha- 2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFNalpha- 2a 180 mcg | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFNalpha- 2a 180 mcg
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/8 | 0/19 | 0/25 | 0/7 | 0/17 | 0/26 | 0/8 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/8 | 0/19 | 0/25 | 0/7 | 0/17 | 0/26 | 0/8 | 1/17
Other Adverse Events (participants affected / at risk) | 19/27 | 8/8 | 15/19 | 21/25 | 7/7 | 13/17 | 15/26 | 5/8 | 11/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+ PegIFN-alpha-2a 180 mcg (N=27) | IP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFNalpha- 2a 180 mcg (N=8) | IP: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFNalpha- 2a 180 mcg (N=19) | CP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg (N=25) | CP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFNalpha- 2a 180 mcg (N=7) | CP: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFNalpha- 2a 180 mcg (N=17) | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg (N=26) | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFNalpha- 2a 180 mcg (N=8) | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFNalpha- 2a 180 mcg (N=17)
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+ PegIFN-alpha-2a 180 mcg (N=27) | IP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFNalpha- 2a 180 mcg (N=8) | IP: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFNalpha- 2a 180 mcg (N=19) | CP: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg (N=25) | CP: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFNalpha- 2a 180 mcg (N=7) | CP: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFNalpha- 2a 180 mcg (N=17) | FU: Cohort 1: JNJ-3989 200 mg+JNJ-6379 250 mg+NA (245/25 mg)+PegIFN-alpha-2a 180 mcg (N=26) | FU: Cohort 1: JNJ-3989 200 mg + NA (245/25 mg) + PegIFNalpha- 2a 180 mcg (N=8) | FU: Cohort 2: JNJ-3989 200 mg + NA (245/25 mg) + PegIFNalpha- 2a 180 mcg (N=17)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 4 | 2 | 0 | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 7 | 2 | 1 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctival Hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye Pruritus (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myopia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Visual Impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0
Aphthous Ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dental Caries (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Food Poisoning (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mouth Ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 2 | 2 | 5 | 2 | 4 | 0 | 1 | 0
Hyperthermia (General disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Influenza Like Illness (General disorders) | 0 | 0 | 0 | 4 | 1 | 2 | 2 | 0 | 1
Injection Site Bruising (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Injection Site Erythema (General disorders) | 0 | 1 | 1 | 3 | 1 | 3 | 0 | 0 | 0
Injection Site Pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection Site Pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection Site Rash (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Injection Site Reaction (General disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Injury Associated with Device (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 1 | 3 | 0 | 3 | 1 | 1 | 1
Temperature Intolerance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Food Allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mite Allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal Allergy (Immune system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspergilloma (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Carbuncle (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 2 | 2 | 4 | 3 | 0 | 0 | 7 | 1 | 0
Hepatitis B (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lower Respiratory Tract Infection Viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 2
Oral Herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory Tract Infection Viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Skin Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 8 | 0 | 1 | 2 | 0 | 4 | 0 | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 2 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood Glucose Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Body Temperature Increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Glucose Urine Present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Liver Scan Abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutrophil Count Decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Ultrasound Liver Abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight Decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
White Blood Cell Count Decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Iron Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 0
Limb Mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 1
Haemangioma of Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Amnestic Disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness Postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 5 | 3 | 2 | 5 | 0 | 1 | 0 | 1 | 1
Neuropathy Peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety Disorder (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Apathy (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed Mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Allergic Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 2 | 1 | 2
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2021-11-25): https://cdn.clinicaltrials.gov/large-docs/39/NCT04439539/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-27): https://cdn.clinicaltrials.gov/large-docs/39/NCT04439539/SAP_001.pdf